CLINICAL TRIAL: NCT05493930
Title: An Easy-to-use Artificial Intelligence Preoperative Lymph Node Metastasis Predictor (LN-MASTER) in Rectal Cancer Based on a Privacy-preserving Computing Platform: Multicenter Retrospective Cohort Study
Brief Title: A Lymph Node Metastasis Predictor (LN-MASTER) in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xishan Wang, Chief of Colorectal Cancer Surgery, Peking Union Medical College
Other Study IDs: XWang
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Rectum Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- development set;: RC patients from the Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College
  Interventions: Other: The hospital where the treatment is performed
- external validation sets 1: RC patients from Changhai Hospital, Naval Medical University
  Interventions: Other: The hospital where the treatment is performed
- external validation sets 2: RC patients from the Second Affiliated Hospital of Harbin Medical University
  Interventions: Other: The hospital where the treatment is performed

INTERVENTIONS:
Other: The hospital where the treatment is performed

SUMMARY:
In this study, we aim to develop and validate an easy-to-use machine learning prediction model to preoperatively identify the lymph node metastasis status for rectal cancer patients by using these clinical data from three hospitals.

DETAILED DESCRIPTION:
In this study, participants were recruited from the Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College (development set), Changhai Hospital, Naval Medical University (external validation set 1), and the Second Affiliated Hospital of Harbin Medical University (external validation set 2), between January 1, 2016, and December 31, 2020. According to the inclusion criteria, participants who (a) were in American Joint Committee on Cancer (AJCC) stages I -III rectal cancer and (b) underwent radical surgery were recruited. In contrast, the exclusion criteria were as follows: (a) other malignancies, (b) received treatment with endoscopic submucosal dissection (ESD), (c) metastatic lesions, (d) did not undergo lymph node dissection, (e) had unavailable assessed lymph node status, and (f) received neoadjuvant therapy. The lymph node metastasis (LNM) status was determined based on the pathological diagnosis of the surgical specimens.

Clinicopathological features included sex, age, body mass index (BMI), comorbidity, distance from the lower edge of the tumor to the anus, carcinoembryonic antigen (CEA) levels, carbohydrate antigen 19-9 (CA19-9) levels, tumor size, degree of tumor differentiation, tumor histology, vascular or lymphatic vessel invasion, AJCC T stage, clinical diagnosis of LNM, and the pathological diagnosis of LNM. Among these, sex, age, BMI, and comorbidities of each participant, such as diabetes, hypertension, hyperlipidemia, and other chronic systemic diseases, were extracted from the electronic hospital information system. Preoperative CEA and CA19-9 levels were obtained from hematological examinations at the time of rectal cancer diagnosis. The distance from the lower edge of the tumor to the anus, differentiation degree, and tumor histology were recorded based on the results of endoscopy and endoscopic biopsies. The tumor diameter and clinical diagnosis of LNM were defined using preoperative pelvic MRI or CT. The diagnosis of vascular invasion, lymphatic vessel invasion, and LNM was based on postoperative pathological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) stages I -III rectal cancer
* underwent radical surgery

Exclusion Criteria:

* other malignancies
* received treatment with endoscopic submucosal dissection (ESD)
* metastatic lesions
* did not undergo lymph node dissection
* had unavailable assessed lymph node status
* received neoadjuvant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: rectal cancer patients with/without lymph node metastasis
Sampling Method: Non-Probability Sample
Enrollment: 6578 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
diagnosis of lymph node metastasis | through study completion, an average of 1 month
  The lymph node metastasis (LNM) status was determined based on the pathological diagnosis of the surgical specimens.

REFERENCES:
- [Derived] Guan X, Yu G, Zhang W, Wen R, Wei R, Jiao S, Zhao Q, Lou Z, Hao L, Liu E, Gao X, Wang G, Zhang W, Wang X. An easy-to-use artificial intelligence preoperative lymph node metastasis predictor (LN-MASTER) in rectal cancer based on a privacy-preserving computing platform: multicenter retrospective cohort study. Int J Surg. 2023 Mar 1;109(3):255-265. doi: 10.1097/JS9.0000000000000067. PMID 36927812